CLINICAL TRIAL: NCT05613309
Title: Clinical Characteristics Analysis and Prediction Model Establishment of Fatal Esophageal and Gastric Variceal Bleeding
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, ChenMingkai, Professor, Renmin Hospital of Wuhan University
Other Study IDs: WDRY2022-K204
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Acute Variceal Bleeding
Keywords: Acute variceal bleeding; Mortality risk prediction model

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with acute varicose hemorrhage in Renmin Hospital of Wuhan University in recent 10 years: In this study, patients with liver cirrhosis and acute variceal bleeding in Renmin Hospital of Wuhan University in the past 10 years will be selected as the research objects. Patients will be divided into survival and death groups according to whether they died 6 hours after admission. The differences in clinical data between the two groups will be compared and analyzed to decide the risk factors for early death and establish a mortality risk prediction model.

SUMMARY:
The purpose of this study is to analyze the clinical characteristics of patients with fatal acute variceal bleeding (AVB) and establish a mortality risk prediction model to identify patients at high risk of death after admission, so as to guide clinical practice, further optimize the allocation of emergency resources, and further reduce the mortality of AVB patients.

DETAILED DESCRIPTION:
How to predict adverse outcomes of acute variceal bleeding and identify high-risk patients remains unclear. Most studies related to risk factors for adverse outcomes in AVB patients took 5 days and 6 weeks as time nodes, and the main outcome indicators were the rebleeding rate and mortality rate at 5 days and 6 weeks. However, some patients admitted to hospital may suffer death within a short period of time ,the investigators will define AVB patients at high risk of death in several hours after admission as fatal acute variceal bleeding.To identify such patients and give more positive treatment can further reduce the mortality of AVB. Such risk stratification can be used to further guide the rational allocation of emergency resources, improve the efficacy of medical resources. This study intends to retrospectively collect the clinical data of AVB patients in Renmin Hospital of Wuhan University, analyze the risk factors for death after admission, establish a mortality risk prediction model, and compare and validate the new model and the scoring model to be verified.

ELIGIBILITY:
Inclusion Criteria:

1. History of cirrhosis/previous history of endoscopic varicose veins/undiagnosed liver disease but signs related to liver disease, hematemesis or melena; The diagnosis of cirrhosis is based on liver biopsy or the usual clinical and radiological criteria;
2. AVB was confirmed by endoscopy without special medical history;

Exclusion Criteria:

1. Patients who cannot obtain complete data (vital signs, medical history, laboratory tests and other data are seriously missing);
2. Patients with upper gastrointestinal bleeding have no evidence of AVB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute varicose hemorrhage in Renmin Hospital of Wuhan University in recent 10 years
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Acute death occurred after admission | Six hours after admission
  Death in patients with acute varicose bleeding in cirrhosis occurs within a short time (initially defined as less than 6 hours after admission)

CONTACTS AND LOCATIONS:
Overall Officials: Mingkai Chen, PHD, Study Director — Renmin Hospital of Wuhan University
Locations (1):
- Mingkai Chen, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided